CLINICAL TRIAL: NCT03811483
Title: Fluid Treatment and the Impact of Gender in a Septic Population
Brief Title: SepsisFLAGS ( FLuidAndGender)
Acronym: FLAGS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christer Svensen, Professor, Karolinska Institutet
Other Study IDs: Sepsis-FluidsandGender
Record Dates: First submitted 2019-01-11; First posted 2019-01-22 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sepsis
Keywords: Fluid Therapy; Gender difference
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female gender
- Male gender

SUMMARY:
In this single-center study the investigators will analyze gender differences among patients with suspected sepsis admitted to the Emergency Department at Södersjukhuset during a period of two years. About 11 000 patients will be included. Patient data including fluid therapy will be drawn from the electronic medical record; Take Care and Clinisoft. In the logistic regression analysis, the investigators will adjust for age, gender, comorbidities, vital signs, preliminary focus of infection, level of care and renal replacement therapy. The aim is to analyze gender differences in fluid treatment and the response to fluid treatment and if the treatment is associated with differences in mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department with suspected sepsis (defined by blood culture taken and intravenous sepsis-antibiotics prescribed within 48 hours) and fulfilling sepsis-3 definition of sepsis (sequential organ failure assesment score of 2 or more)

Exclusion Criteria:

* Patients transferred from other hospitals or treatment clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is patients admitted at the emergency department at Södersjukhuset in Southern Stockholm. Södersjukhuset has 600 hospital beds and manages most medical fields except for highly specialized care for example neuro and thoracic surgery. 130 000 patients are seeking medical care yearly which makes the emergency department at Södersjukhuset the most frequented in Scandinavia.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Gender differences in fluid treatment | Fluid therapy during the first six hours (adherence to sepsis bundles) and the first five days after admission.
  Millilitres of fluid given per kilogram of patient weight (ml/kg).

SECONDARY OUTCOMES:
Association between amount of fluid and mortality | In-Hospital Mortality, 30- and 90-days mortality
  Analyze the whole cohort and female/ male gender as subgroups
Type of fluids | First five days after admission.
  Type according to Anatomical, Therapeutic and Chemical Classification System
Association between fluid therapy and levels of lactat | First five days efter admission
  Analyze the whole cohort and female/ male gender as subgroups
Association between fluid therapy and need for/ dose of vasopressors/inotropic drugs | First five days efter admission
  Analyze the whole cohort and female/ male gender as subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jonmarker, Principal Investigator — Karolinska Institutet, Södersjukhuset
Locations (1):
- Södersjukhuset, Stockholm, Stockholm County, Sweden